CLINICAL TRIAL: NCT01261286
Title: Pharmacodynamics and Pharmacokinetics of Verapamil in Crohn's Disease Patients
Brief Title: Drug-Disease Interaction in Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Dr. Richard Fedorak, University of Alberta
Other Study IDs: VER-2010
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Crohn's Disease
Keywords: inflammation; receptor downregulation; reduced response; calcium channels; PK-PD relationship
MeSH Terms: conditions — Crohn Disease; Inflammation | interventions — Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: verapamil

SUMMARY:
Objective: To determine the effect of C-reactive protein (CRP) status, and infliximab treatment on the pharmacodynamics and pharmacokinetics of verapamil, a model drug for L-type calcium channel blocking, in Crohn's disease (CD) patients compared to healthy patients.

Hypotheses:CD patients will have elevated plasma verapamil concentrations, but diminished dromotropic response to verapamil; the concentration of circulating norepinephrine, used as a surrogate marker of sympathetic nervous activity, will be similar between the healthy patients and the CD patients; the sympathetic nervous system of the heart will be similar to healthy patients; Crohn's disease patients with normal CRP will have higher drug response compared to high CRP (>3 mg/l) patients; and that infliximab-treated patients will have higher verapamil response than those with similar symptom profiles who are not infliximab treated.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to adhere the study protocol
* Males of females of non-childbearing potential aged from 18 to 65 years
* Lab values no more than 10% outside of the lab's stated normal range unless the subject is in the Crohn's disease group and the values are related to the disease, or if the PI decides the abnormality is not clinically significant
* The subject is healthy (except for the Crohn's disease group)
* Non-smoker for at least 3 months

Exclusion Criteria:

* History of hypersensitivity to verapamil
* Significant history of gastrointestinal (other than Crohn's disease), liver, kidney, or any other disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
* Significant history of allergies
* Significant history of cardiovascular or hematological disease
* Significant history of asthma, chronic bronchitis or bronchospastic conditions
* Presence of diabetes mellitus or any other condition which would preclude fasting
* Maintenance therapy with any drug (except those prescribed for Crohn's disease) or a history of drug dependence, alcohol abuse, or serious psychological disease
* Any clinically significant illness other than Crohn's disease in the previous 30 days prior to the study
* Use of enzyme-modifying drugs in the previous 30 days before the study
* Blood donation in the previous 56 days or multiple blood samplings in the previous 30 days before the study
* History of fainting upon blood sampling
* Participation in another clinical trial within 30 days of the study
* Narcotic use
* Glucocorticoid treatment in the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Richard Fedorak, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada